CLINICAL TRIAL: NCT05034289
Title: Reducing Racial Disparities in Cancer Care With PINPOINT (Promoting INformed Approaches in Precision Oncology and ImmuNoTherapy)
Brief Title: Promoting INformed Approaches in Precision Oncology and ImmuNoTherapy
Acronym: PINPOINT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: American Cancer Society, Inc. (Other); Pfizer (Industry)
Responsible Party: Principal Investigator, Anita Y. Kinney, PhD, RN, Study Principal Investigator; Associate Director for Cancer Health Equity, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 132101; Pro2021000072 (Other: Rutgers, The State University of New Jersey)
Record Dates: First submitted 2021-08-27; First posted 2021-09-05 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Clinical Trials; Immunotherapy

STUDY DESIGN:
Intervention Model Description: A community-engaged approach, including a Community Advisory Board and two rounds of key informant interviews with Black patients with cancer, their relatives, and providers (n = 48) were used to develop and refine the multimedia digital intervention. Thematic analysis was conducted for qualitative data. The intervention was then pilot-tested with 33 Black patients with cancer to assess feasibility, acceptability, appropriateness, knowledge, decision self-efficacy, and patient empowerment; Wilcoxon matched-pairs signed-rank test was used to analyze quantitative data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PINPOINT Digital Educational Tool (Experimental): Newly diagnosed Black cancer patients will be asked to access and engage with the educational website/intervention prototype before their clinic visit or in the clinic immediately before their appointment with their treating oncologist.
  Interventions: Behavioral: PINPOINT Digital Educational Tool

INTERVENTIONS:
Behavioral: PINPOINT Digital Educational Tool — The intervention prototype called the PINPOINT Digital Educational Tool will be comprised of four main sections that include information about: 1) precision oncology; 2) clinical trials; 3) "Learn More" screens; and 4) discussion points and questions for the treating clinician. The intervention prototype will also include a search function, short videos of patient testimonials, patient-provider interaction about immunotherapy and clinical trials, as well as a list of questions/concerns that the patient could print (or save electronically) and take with them to their provider visit. An optional chatbot will be available in the corner of the screen. Users can ask the chatbot questions about any of the material on the website or request additional information. The chatbot will also be able to help patients search for molecularly targeted and immunotherapy clinical trials and offer additional resources (such as websites and online support groups).

SUMMARY:
The purpose of the research is to: develop an educational website to empower Black and African American cancer patients to make informed decisions about personalized cancer treatment and clinical trials. The sample size for the qualitative interviews was (n=48) when saturation was achieved. With a goal of (n=33) for the pilot trial, the overall target sample size for the study is (n=81).

DETAILED DESCRIPTION:
The website offers tools for discussing innovative treatments with their clinicians, finding clinical trials, and locating support groups. We are conducting key informant interviews, testing the website with pilot tester and asking volunteers from our Community Advisory Board to review our website prototype to further improve its design and features.

ELIGIBILITY:
Inclusion Criteria

Patient Key Informant:

* Age 18 and older
* Self-identify as Black/African American
* Diagnosed with solid tumor
* Able to read and speak English fluently
* Able to provide informed consent
* Able to complete 1 survey and an in-depth interview

Relative Key Informant:

* Age 18 and older
* Spouse, blood relative, or caregiver of a cancer patient who identifies as Black/African American
* Able to read and speak English fluently
* Able to provide informed consent
* Able to complete 1 survey and an in-depth interview

Provider Key Informant:

* Age 18 and older
* Physician, nurse, social worker, patient navigator, or financial counselor
* Work in oncology setting
* Able to read and speak English fluently
* Able to provide informed consent
* Able to complete 1 survey and an in-depth interview

Pilot Tester:

* Age 18 and older
* Self-identify as Black/African American
* Able to read and speak English fluently
* Able to provide informed consent
* Newly diagnosed with solid tumor cancer (Stage I-IV)
* Have not yet consulted with an oncologist regarding treatment
* Able to complete 2 surveys and an in-depth interview

Exclusion Criteria

Key informants will be excluded from the study if they do not meet the inclusion criteria. Pilot testers will be excluded from the study if they previously participated as key informants and do not meet inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2023-05-19 (Actual); Study Completion 2023-05-19 (Actual)

PRIMARY OUTCOMES:
Community Advisory Board, Key Informants and Pilot Testers | June 2021-June 2022
  Employ a community-engaged approach, including a Community Advisory Board and key informant interviews, to a) assess knowledge, attitudes, beliefs, and sociocultural, clinical, and system-level factors (e.g., barriers) that may explain disparities in decisions about use of precision oncology in Black cancer patients
Website Development | June 2021-June 2023
  Utilize this information to guide the iterative development and pilot testing of an innovative, patient-centered and culturally tailored internet-based education and decision support intervention, "Promoting INformed approaches in Precision Oncology and ImmuNoTherapy (PINPOINT)," to reduce racial disparities in access to and use of guideline-based therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Y Kinney, PhD, RN, Principal Investigator — Rutgers Cancer Institute
Locations (1):
- The Rutgers Cancer Institute, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2025-07-07): https://cdn.clinicaltrials.gov/large-docs/89/NCT05034289/Prot_001.pdf
  • Informed Consent Form (2025-07-07): https://cdn.clinicaltrials.gov/large-docs/89/NCT05034289/ICF_002.pdf